CLINICAL TRIAL: NCT04494178
Title: A Randomized, Placebo-controlled, Double-blind, Cross-over Study to Evaluate the Effect of G-PUR® on Dietary Fumonisin Bioavailability
Brief Title: G-PUR® for Reduced Dietary Fumonisin Bioavailability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Several analytical laboratories failed to develop and validate a suitable assay of urine fumonisin (the primary endpoint) up to date. Because of missing alternatives for an analytical laboratory the objective of the study cannot be met.
Sponsor: Glock Health, Science and Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: G-Fum_01
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Reduction of Dietary Fumonisin Bioavailability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.0g G-PUR® oral - Placebo (Experimental)
  Interventions: Device: 2.0g G-PUR®; Other: Placebo
- Placebo - 2.0g G-PUR® oral (Experimental)
  Interventions: Device: 2.0g G-PUR®; Other: Placebo

INTERVENTIONS:
Device: 2.0g G-PUR® — Oral administration (Intervention period I)
  Arms: 2.0g G-PUR® oral - Placebo
Device: 2.0g G-PUR® — Oral administration (Intervention period II)
  Arms: Placebo - 2.0g G-PUR® oral
Other: Placebo — Intervention period I
  Arms: Placebo - 2.0g G-PUR® oral
Other: Placebo — Intervention period II
  Arms: 2.0g G-PUR® oral - Placebo

SUMMARY:
This prospective, placebo-controlled, randomized, monocentric, double-blind, crossover study in healthy volunteers aims to assess the effect of a single dose of 2 g G-PUR® on bioavailability of dietary fumonisin and to evaluate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects
2. Age 18-55 years
3. BMI 17-27
4. Subjects are in good clinical and mental health as established by medical history and physical examination
5. Subject understands the scope of the study and agrees to strictly adhere to the study related diet plan
6. Written informed consent

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Lack of willingness or capacity to co-operate appropriately
3. Regular use of medications in the previous 2 months (except oral contraception)
4. History of malignancies within the past two years or on current anticancer treatment
5. History of gastrointestinal pathology such as clinically relevant gastritis, gastric ulcers, inflammatory bowel disease, chronic constipation
6. History of diarrhoea within the past 14 days of screening
7. History of gastrointestinal surgery with exception of appendectomy
8. History of any chronic liver disease
9. History of autoimmune disease requiring treatment within the past two months of screening
10. Known symptomatic food allergies
11. Active infection (including HIV and hepatitis B or C), or abnormalities in laboratory testing, vital signs, or physical examination
12. Hypersensitivity to aluminium and/or silicon
13. Chronic renal disease requiring dialysis
14. Alcohol, cigarette or drug abuse
15. Presence of any condition that impacts compliance with the study procedures
16. Use of any investigational or non-registered product (drug or device) within 30 days preceding the first study product administration, or planned use during the study period
17. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse) or relationship to the sponsor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
The bioavailability of fumonisin is estimated based on the concentration of urinary biomarkers FB1 and FB2 | 24 hours

SECONDARY OUTCOMES:
Incidence of (serious) adverse device effects | 19 days
Urinary biomarkers FB1 and FB2 (separately and sum of FB1 and FB2) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof.Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria